CLINICAL TRIAL: NCT04845061
Title: Evaluating the Outcome of Cardio Selective beta1- Blockers Use in Patients With Chronic Obstructive Pulmonary Disease: A Pilot Study
Brief Title: Evaluating the Outcome of Cardio Selective beta1- Blockers Use in Patients With Copd
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Asma Shain Suliman, Clinical pharmacist, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: beta blockers in copd
Record Dates: First submitted 2021-03-29; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Copd
Keywords: beta blockers -nebivolol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nebivolol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nebivolol then placebo (Placebo Comparator): Comprises15 copd patients, after recruitment in study and written informed consent, patient's administered nebivolol (1.25 mg for one week then2.5mg fore another one week and 5 mg at 8am for 10 weeks)and washout period4 weeks then shifted to placebo for 12 weeks
  Interventions: Drug: Nebivolol Tablets
- placebo then nebivolol (Active Comparator): Contain 15 copd patient's after recruitment and Written informed consent administered placebo for 12 weeks and washout period for 4 weeks then shifted to nebivolol for 12 weeks
  Interventions: Drug: Nebivolol Tablets

INTERVENTIONS:
Drug: Nebivolol Tablets — cardio selective beta-1 blocker

SUMMARY:
To Evaluate the Outcome of cardio selective beta1 (β1-) blockers use in patients with chronic obstructive pulmonary disease.

Patient education about the COPD and their medications.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common preventable and Treatable airway disorder characterized by symptoms such as dyspnea, chronic Cough, and sputum production along with persistent airflow limitation that is not fully Reversible.

Evidence provided by post hoc analysis of clinical trials and large observational studies suggests a beneficial effect of beta-blockers on mortality and exacerbation in mild to moderate COPD patients.

Evidence concerning cardio selective B blockers. Over the past 20 years' non selective B blockers have largely been replaced with cardio selective blockers. Cardio selective beta blockers such as atenolol and metoprolol are at least 20 times more potent at blocking B-1 receptors than B-2 receptors. At therapeutic doses the B-1 blocking effect, and therefore the risk of bronco constriction, is negligible. In addition there is strong evidence that B-blocked cause up-regulation and sensitization of B-receptors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. informed consent.
3. Age >40years.
4. FEVl/FVC<70%.
5. diagnosed 3 month before enrollment (mild-moderate)
6. Reversability test pre-post bronchodilators FEVl predicted<200ml/hr and less than 12%.

Exclusion Criteria:

1. Asthmatic patient.
2. patient already use B blockers.
3. Acute exacerbation.
4. Pregnency -lactation.
5. Advanced cardiac, renal or liver disease according to investigator opinion.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
forced vital capacity | 3 months
  amount of air that can be forcibly exhaled from the lung after taking the deepest breath possible (FVC\liter)
forced expiratory volume in one second | 3 month
  volume of air exhaled under condition in the first second (FEV1\liter)
blood pressure | 3 month
  BP millimetre mercury

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Chest Department, Ain Shams University Hospitals, Cairo, Egypt., Cairo
  - Chest Department, Ain Shams University Hospitals, Cairo

IPD SHARING:
Plan to Share IPD: Undecided